CLINICAL TRIAL: NCT00966745
Title: Effect of Milrinone During Living Donor Hepatectomy Using a Low Central Venous Pressure Technique
Brief Title: Milrinone During Living Donor Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mil_living_liver_donor
Record Dates: First submitted 2009-08-13; First posted 2009-08-27 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-08

CONDITIONS: Hepatectomy
Keywords: surgical field condition
MeSH Terms: interventions — Milrinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- milrinone (Active Comparator): milrinone infusion
  Interventions: Drug: milrinone
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: milrinone
  Arms: milrinone
Drug: placebo
  Arms: placebo

SUMMARY:
Maintaining a low central venous pressure during living donor hepatectomy is routine practice. The investigators tried to test the hypothesis that using milrinone to maintain a low central venous pressure (CVP) during is associated with a superior surgical field and less blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Living liver donors

Exclusion Criteria:

* Donors with concurrent cardiac, pulmonary, and urologic disease
* Hepatectomy performed laparoscopically

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
condition of surgical field | intraoperative period (from the start of surgery to end of living donor hepatectomy)

SECONDARY OUTCOMES:
the use of vasopressor and diuretics to maintain hemodynamic stability and low CVP status, respectively | intraoperative period (from the start of surgery to end of living donor hepatectomy)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea